CLINICAL TRIAL: NCT02527590
Title: Development of Stimulator Pneumatic for Realization of Evoked Potential Allodynic/Somatosensory
Acronym: STIMEA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1008057; 2010-A00568-31 (Other: AFSAPPS)
Record Dates: First submitted 2015-08-11; First posted 2015-08-19 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2016-08

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient with neuropathic pain with allodynia (Experimental)
  Interventions: Other: pneumatic stimulations(allodynic area); Other: pneumatic stimulations (healthy area); Other: no stimulation (control)
- healthy volunteers (Experimental)
  Interventions: Other: pneumatic stimulations no auditory masking; Other: no stimulation (control); Other: pneumatic stimulations with audidory masking

INTERVENTIONS:
Other: pneumatic stimulations(allodynic area) — 2 series of 20 pneumatic stimulations (air jet) on a allodynic area for recording evoked potentials
  Arms: patient with neuropathic pain with allodynia
Other: pneumatic stimulations (healthy area) — 2 series of 20 pneumatic stimulation on a healthy area (either contralateral or above or below allodynic area) will no pain triggering for recording evoked potentials
  Arms: patient with neuropathic pain with allodynia
Other: pneumatic stimulations no auditory masking — 2 series of pneumatic stimulations (air jet) on the hand (without feeling pain) for recording evoked potentials
  Arms: healthy volunteers
Other: no stimulation (control) — no stimulation (control condition): air jet directed beside the hand
Other: pneumatic stimulations with audidory masking — 2 series of 20 pneumatic stimulations (air jet) on the hand (without feeling pain) with auditory helmet that totally masked the air jet noise.
  Arms: healthy volunteers

SUMMARY:
The stimuli used in the evoked potentials are electrical or laser. They are started and synchronized with the collection of the EEG by signals TTL (transistor-transistor logic). Investigators propose to validate a pneumatic stimulator delivering the compressed air sync with the EEG. It has two advantages over existing stimuli: Is capable of inducing in patients an allodynic response, excessive, painful, in response to a stimulation painless rarely obtained with laser or electrical stimuli. Therefore, the pneumatic stimulation is a means to study allodynic evoked potentials unknown to date.

It must be possible with a single stimulator to explore non-painful sensations and allodynic sensation , compare them with one device. The differences are the abnormal responses. This validation assumes evoked potential recording 1. somatosensory (low stimulation) then 2. allodynic (only in patients). The study therefore provides for the registration 100 potential for each of these two modalities in patients and only for the painless pneumatic modality in volunteers.

ELIGIBILITY:
Inclusion Criteria of patients :

* Major Patient
* Patient affiliated or entitled to a social security scheme
* Patient with neuropathic pain authenticated by the neurologist, with the presence of allodynia.
* Patient has given its written consent to participate in the study

Exclusion Criteria of patients :

* Diseases affecting the nervous system,
* Diabetes,
* Patients who received chemotherapy
* Pregnant woman
* Nobody in emergencies
* A person unable to give consent

Inclusion Criteria of healthy volunteers :

* Major subject
* Subject affiliated or entitled to a social security scheme
* Subject has given its consent to participate in the study

Exclusion Criteria of healthy volunteers :

* Diseases affecting the nervous system,
* Diabetes,
* Patients who received chemotherapy
* Pregnant woman
* Nobody in emergencies
* A person unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
composite outcomes : latencies and amplitudes of pneumatic evoked potential | Day 1
  latencies (in ms) and peak-to-peak amplitudes (in μV) were measured on the electrode providing the response with the highest amplitude.

SECONDARY OUTCOMES:
latencies evoked potentials allodynic tires | Day 1
  The latencies of allodynic evoked potentials (allodynic patients) and latencies of somesthetic evoked potentials (healthy volunteers). The mean of latencies somatosensory evoked potentials in healthy volunteers will be calculated with its confidence interval. Thus, for each patient allodynic if the latency of its response is not included in this confidence interval then his answer will be considered pathological.

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No